CLINICAL TRIAL: NCT01716611
Title: Efficacy and Safety Study of Tolvaptan for Liver Cirrhotic Patients With Hyponatremia and Ascites: A Multi-center, Randomized, Double-blind, Placebo-controlled 4-weeks Clinical Trial
Brief Title: Tolvaptan for Hyponatremia in Cirrhotic Patients With Ascites
Acronym: TONIC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Konkuk University Medical Center (Other)
Collaborators: Inje University (Other); Korea University Anam Hospital (Other); Hanyang University (Other); Severance Hospital (Other); Seoul St. Mary's Hospital (Other); Samsung Medical Center (Other); Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); Hallym University Medical Center (Other); Inha University Hospital (Other); Soonchunhyang University Hospital (Other); Kyungpook National University Hospital (Other); Incheon St.Mary's Hospital (Other); Chungnam National University (Other)
Responsible Party: Principal Investigator, Won Hyeok Choe, Associate Professor, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KUH1010412
Record Dates: First submitted 2012-10-18; First posted 2012-10-30 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Hyponatremia; Ascites
Keywords: liver cirrhosis; hyponatemia; ascites; vaptans; antidiuretic hormon; arginine vasopressin
MeSH Terms: conditions — Hyponatremia; Ascites; Liver Cirrhosis; Diabetes Insipidus | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tolvaptan group (Active Comparator): Form : Tablet, Dosage: 15 mg, 30 mg or 60 mg, Frequency: once a day. Duration: 28days
  Interventions: Drug: Tolvaptan
- Placebo group (Placebo Comparator): Form : Tablet, Dosage: 15 mg, 30 mg or 60 mg, Frequency: once a day. Duration: 28days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Tolvaptan — 15 - 60 mg/day for 28 days
  Other Names: SAMSCA
  Arms: Tolvaptan group
Drug: placebo
  Arms: Placebo group

SUMMARY:
The purpose of the study is to investigate the efficacy and safety for the management of hyponatremia and ascites in patients with liver cirrhosis.

DETAILED DESCRIPTION:
Patients with advanced cirrhosis frequently develop dilutional hyponatremia due to impairment of their renal ability to eliminate solute-free water. Although the pathophysiology of this disorder is multifactorial, an increased hypersecretion of arginine vasopressin (AVP) is a major factor. The prevalence of hyponatremia in cirrhosis, as defined by a serum sodium level of 130 mmol/L is reported to be about 20%, and there are several lines of evidence that hyponatremia is a risk factor for the development of hepatic encephalopathy, and that it predicts a poor quality of life independent of liver function. Hyponatremia also predicts short-term mortality in cirrhotic patients awaiting liver transplantation. The principle of the management of hypervolemic hypona- tremia is to induce a negative water balance, with the aim of normalizing the increased total body water, which would result in an improvement in serum sodium concentration. Fluid restriction is the most widely accepted nonpharmacological therapy, but its efficacy is very limited. The administration of hypertonic sodium chloride has been common in severe hypervolemic hyponatremia, but its effect is only partial and short lived; moreover, additional expansion of fluid can worsen ascites and edema. Therefore, the pathophysiologically oriented treatment of hyponatremia focuses on inhibiting the actions of AVP. Recently, antagonists of the V2 receptors of vasopressin has been proposed to manage hyponatremic patients, such as heart fauilure, syndrome of inappropriate antidiuretic hormone or liver cirrhosis. Especially, a lot of hyponatremic patients with cirrhosis had ascites, and some of them had intractable ascites. In these patients, antagonists of the V2 receptors of vasopressin including tolvaptan might have beneficial effect in enhancing not only hyponatremia , but also ascites

ELIGIBILITY:
Inclusion Criteria:

1. 20 years of age or older
2. Patients with cirrhosis as diagnosed by liver biopsy or a combination of laboratory (thrombocytopenia), radiologic (cirrhotic feature of liver, splenomegaly, collateral shunt on US, CT, or MRI) and endoscopic findings (gastoesophageal varices or portal hypertensive gastropathy)
3. ≥ Grade 2 ascites who have already been treated with restricted salt diet within 3 month
4. Hyponatremia (Serum sodium ≥120 mEq/L and ≤130 mEq/L)
5. Written informed consent

Exclusion Criteria:

1. Hypovolemic hyponatremia (Patients with hypotension or chronic heart failure)
2. Serum potassium concentration > 5.5 mEq/L
3. Serum bilirubin > 5.0 mg/dL
4. Blood coagulation factor < 40% or international normalized ratio (INR) > 2.3
5. Platelet count < 30,000/mm3
6. Serum creatinine > 3 mg/dL
7. Treatment within 2 weeks with vasopressin anlogues
8. Systolic blood pressure <80 mmHg
9. History of gastrointestinalesophageal varix bleeding variceal hemorrhage
10. Spontaneous bacterial peritonitis
11. Hepatic encephalopathy ≥ grade 3
12. History of Hepatocellular carcinoma treatment within 3month or viable tumor Viable hepatocellular carcinoma
13. Liver transplant
14. Previous treatment with transjugular intrahepatic portosystemic stent shunt (TIPS)
15. History of significant cardiac diseases such as recent myocardial infarction or ischemic diseases within 1 year of screening
16. Prolonged QTc interval of > 500 ms based on electrocardiography
17. Treatment within 2 weeks with substances or drugs that may either induce or significantly inhibit cytochrome P450 3A (ketoconazole, clarithromycin, erythromycin, fluconazole, diltiazem, verapamil, etc)
18. Pregnant or breast feeding
19. Patients with galactose intolerance or malabsorption (as production of the drug contains lactose)
20. HbA1Cc ≥ 9 %
21. Serious medical illness (e.g. heart failure, severe pulmonary disorders, alcohol dependence, malignant tumors, etc)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-01 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
the change in the average daily area under the curve (AUC) for the serum sodium concentration from baseline to day 28 after intervention | baseline and 28 days

SECONDARY OUTCOMES:
the change in the average daily area under the curve (AUC) for the serum sodium concentration from baseline to day 4 | baseline and 4 days
the time to normalization of the serum sodium concentration | up to 28 days
the time to first paracentesis, number of paracentesis, the volume of ascitic fluid obtained from paracentesis | up to 28 days
Abdominal discomfort based on a 100-mm visual analogue scales (VAS) | day 1, 2, 3, 4, 7, 14, 21, 28
The change in the dose of concomitant diuretics from baseline at day 28 | day 1, 2, 3, 4, 7, 14, 21, 28
the number of participants with serious adverse events | from baseline to day 28 after intervention
the time to ascites improvement | up to 28 days
the time of worsening of ascites | up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: June Sung Lee, MD, PhD, Principal Investigator — Inje University Ilsan Paik Hospital
Locations (1):
- Konkuk University Medical Center, Seoul, Seoul, South Korea